CLINICAL TRIAL: NCT01602601
Title: A Study to Test the Possibility of Cross Reaction of the Antibodies Induced by the ELAPRASE (R) to GSK2788723 ELAPRASE is a Trade Mark Owned by a Third Party
Brief Title: A Study to Test the Possibility of Cross Reaction Induced by the Idursulfase Drug to GSK2788723
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116406
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Mucopolysaccharidosis II
Keywords: Hunter syndrome, immunogenicity, antibodies
MeSH Terms: conditions — Mucopolysaccharidosis II | interventions — idursulfase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples will be collected and serum will be analyzed and retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Patients will have a single blood draw for the analysis of antibodies induced by idursulfase. Samples will be used to further evaluate whether the antibodies induced by idursulfase bind to GSK2788723 molecules in vitro and if these antibodies neutralize the bioactivity of GSK2788723 in vitro.
  Interventions: Drug: Idursulfase; Drug: GSK2788723

INTERVENTIONS:
Drug: Idursulfase — recombinant version of IDS produced from human fibroblast. idursulfase is approved for every week (EW) intravenous (IV) administration.
  Other Names: recombinant IDS
Drug: GSK2788723 — GSK2788723 is being developed by JCR and GSK for the treatment of Hunter syndrome

SUMMARY:
Study IDS116406 will be a non-interventional, phlebotomy study in Hunter Syndrome patients who are currently being treated with idursulfase, an enzyme replacement therapy, and in at least a single patient who is naïve to treatment, if possible to recruit. All patients enrolled into the study will have a single blood draw for the analysis of antibodies induced by this enzyme replacement therapy (idursulfase). Patient samples with positive responses to antibodies induced by idursulfase will be used to further evaluate whether the antibodies induced by idursulfase bind to GSK2788723 molecules in vitro and if these antibodies neutralize the bioactivity of GSK2788723 in vitro. Each subject will have a screening visit, which may occur at their regularly scheduled out-patient visit. If the patient consents to participate in the study, a blood sample (total volume of approximately 3mL) for immunogenicity analysis will be drawn before their current treatment infusion

DETAILED DESCRIPTION:
Study IDS116406 will be a non-interventional, phlebotomy study in Hunter Syndrome patients who are currently being treated with idursulfase, an enzyme replacement therapy, and in at least a single patient who is naïve to treatment, if possible to recruit. All patients enrolled into the study will have a single blood draw for the analysis of antibodies induced by this enzyme replacement therapy (idursulfase). Patient samples with positive responses to antibodies induced by idursulfase will be used to further evaluate whether the antibodies induced by idursulfase bind to GSK2788723 molecules in vitro and if these antibodies neutralize the bioactivity of GSK2788723 in vitro. Each subject will have a screening visit, which may occur at their regularly scheduled out-patient visit. If the patient consents to participate in the study, a blood sample (total volume of approximately 3mL) for immunogenicity analysis will be drawn before their current treatment infusion

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if patient meets criteria 1 and 2 or 1 and 3:

* Diagnosed with Hunter syndrome
* Patients with Hunter syndrome who are being treated with idursulfase
* Patients with Hunter syndrome who are naïve of idursulfase treatment (if possible*) *This study will also attempt to recruit 1 patient who has never received idursulfase. If a naïve patient has not been identified within an agreed amount of time between GSK and the investigator, the study will concluded without this sample

Exclusion Criteria:

* Subjects who are currently participating in another clinical trial are not permitted to be enrolled in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 11 subjects will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-04-09 (Actual); Primary Completion 2012-06-11 (Actual); Study Completion 2012-06-11 (Actual)

PRIMARY OUTCOMES:
Level and capability of binding and neutralizing antibodies induced by idursulfase after the administration of idursulfase | 1 Day
  To assess the cross-reactivity of the antibodies induced by idursulfase to GSK2788723, in vitro

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Results for study 116406 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116406?search=study&search_terms=116406#rs